CLINICAL TRIAL: NCT01548053
Title: A Study Evaluating the Effects of a Primary Care - Dementia Assessment Treatment Algorithm on the Quality of Care Provided to Older Adults With Dementia in Primary Care Settings
Brief Title: The Primary Care - Dementia Assessment and Treatment Algorithm
Acronym: PC-DATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Dallas Seitz, Assistant Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: PC-DATA1
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: Primary care; Dementia; Knowledge translation; Quality of care; Qualitative methods; Alzheimer's disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PC-DATA tool — The implementation plan consists of educational sessions and a dementia care manager (DCM). The educational sessions consist of two components: a 1.5 hour group-based DATA tool implementation workshop with primary care providers (PCPs); and, a 1 hour follow-up session at study mid-point. The DCM will facilitate application of the DATA tool and provide direct support to PCPs during the study.

SUMMARY:
Alzheimer's disease (AD) and related forms of dementia currently affect over 400,000 individuals in Canada and the numbers of community dwelling older adults with AD is rapidly growing. AD is associated with over $15 billion annually in care costs. Most individuals with AD are under the care of primary care providers (PCPs) including family physicians and primary care nurses. The evaluation and management of AD is challenging for PCPs and the quality of care provided to older adults with AD by PCP could be improved which would optimize outcomes for this vulnerable population. Provision of quality care to older adults with AD involves implementation of best practices as outlined in guidelines such as the Canadian Consensus Conference Guidelines on the Diagnosis and Treatment of Dementia. Utilizing a group of dementia researchers, PCPs, other knowledge users, and individuals affected by AD, this project will develop practical, clinically relevant resources for primary care physicians and nurses to aid in the evaluation of older adults with AD. A knowledge tool, the Primary Care - Dementia Assessment and Treatment Algorithm (DATA Tool) will be introduced into several primary care settings in Ontario using educational sessions with PCP with additional support from internet resource and a dementia care manager. The quality of dementia care provided to older adults newly diagnosed with AD will be assessed in the three years preceding the intervention compared to the year following the implementation. This project will also describe the process of knowledge exchange with PCPs, including potential barriers and facilitators of knowledge uptake and examine if the care provided during the intervention was patient-centred through interviews with patients and caregivers.

Research Objectives:

1. Develop knowledge tools to facilitate assessment and treatment of AD by PCPs based on best evidence;
2. Transfer these knowledge tools into a variety of primary care settings in Ontario; and,
3. Evaluate the effects of this intervention on dementia quality of care, PCP application of knowledge, and the patient-centeredness of care.

ELIGIBILITY:
Primary Care Provider Inclusion Criteria:

* Primary care provider at participating sites

Primary Care Provider Exclusion Criteria:

* primary care provider at non-participating site

Patient Inclusion Criteria:

* Community-dwelling at time of initial presentation to primary care provider
* Age 60 years or older at time of initial assessment by primary care provider
* Presenting to primary care providers with cognitive or functional symptoms suggestive of Alzheimer's disease or other form of dementia
* Patient must have a caregiver or substitute decision maker

Patient Exclusion Criteria:

* Prevalent cases of dementia will be excluded from study population
* Individuals with dementia residing in long-term care or nursing homes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in number of dementia care process quality indicators achieved. | 1 year following implementation
  The evaluation of quality indicators (QI) using chart audit data will be undertaken following initial assessment of dementia will be used to assess the quality of care provided to individuals with dementia. The change in number of QI satisfied following the intervention will be compared to a historical group of individuals assessed for dementia by each PCP in the 3 years preceding the intervention.

SECONDARY OUTCOMES:
Impact on learning and knowledge application | Approximately 9 months following intervention
  Qualitative interviews with family physicians and interprofessional primary care professional will be conducted using a grounded theory design will be conducted with primary care providers to identify key conceptual, contextual and process elements involved in the exchange and application of dementia-specific knowledge in the primary care context.
Client-centred care | Approximately 9 months following intervention
  Interviews will be conducted with patients and careviers to seek to identify key elements of patient-centred care.

CONTACTS AND LOCATIONS:
Overall Officials: Dallas P Seitz, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada